CLINICAL TRIAL: NCT00524121
Title: Phase II Study of Erlotinib (Tarceva®) and Radiotherapy for Elderly Patients With Esophageal Carcinoma
Brief Title: Erlotinib and Radiation Therapy in Treating Older Patients With Stage I, Stage II, Stage III, or Stage IV Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563268; RPCI-I-62705 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Erlotinib Hydrochloride; Immunohistochemistry; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Erlotinib (Experimental): Patients receive oral erlotinib hydrochloride once daily for 1 year
  Interventions: Drug: erlotinib hydrochloride; Other: immunohistochemistry staining method; Radiation: radiation therapy

INTERVENTIONS:
Drug: erlotinib hydrochloride — Oral
Other: immunohistochemistry staining method — Correlative Study
Radiation: radiation therapy — Radiation Treatment

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving erlotinib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving erlotinib together with radiation therapy works in treating older patients with stage I, stage II, stage III, or stage IV esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the overall survival of older patients with stage I-IV squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction treated with erlotinib hydrochloride in combination with radiotherapy.

Secondary

* Assess the proportion of patients achieving mucosal complete response after treatment with this regimen.
* Determine the progression-free survival of patients treated with this regimen.
* Assess the effect of this regimen on dysphagia control, performance status, and overall quality of life of these patients.
* Investigate the correlation between smoking status and overall survival of these patients.
* To correlate the Epidermal growth factor receptor (EGFR) and phosphor Epidermal growth factor receptor (pEGFR) expression by IHC and EGFR mutation status with clinical outcomes.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily for 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo external beam radiotherapy 5 days a week in weeks 1-4 or 5 days a week for the first 5.5 weeks.

Tumor tissue samples are analyzed by IHC for the expression of E-cadherin, P-cadherin, vimentin, cytokeratin, phospho-S6, and Ki67.

After completion of study treatment, patients are followed at 30 days and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven primary squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal (GE) junction

  * GE junction tumors with 50% or more tumor located in the esophagus determined by radiologic or endoscopic evaluation
  * Stage I-IVA disease determined by CT scan or MRI of the chest and abdomen

    * Stage IVB disease allowed if metastases to distant regional lymph nodes (celiac or cervical) only and no other sites
* Not a surgical candidate and ineligible for chemotherapy due to any of the following:

  * Neuropathy
  * Cardiac disease
  * Performance status 2
  * General overall condition felt by the investigator to be a contraindication to platinum-based therapy
* Bronchoscopy with biopsy and cytology required if primary esophageal cancer is < 26 cm from incisors
* No evidence of clinically active interstitial lung disease (patients who are asymptomatic with chronic, stable, radiographic lung changes allowed)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 4 months
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin ≤ 1.3 mg/dL
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* No prior malignancies except basal cell or squamous cell skin cancer, in situ cervical cancer, or superficial transitional cell bladder cancer, unless diagnosed and/or treated > 2 years prior to current study and are without evidence of recurrence
* No history of allergy to erlotinib or any of its excipients
* No serious, uncontrolled, concurrent infection
* No clinically serious, uncontrolled medical conditions that the investigator feels might compromise study participation
* No lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* No unwillingness to participate or inability to comply with the protocol for the duration of the study

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for this tumor
* No prior resection or attempted resection of esophageal cancer
* No prior anti-epidermal growth factor receptor therapy (unless given in an adjuvant setting and completed at least 12 months earlier)
* No participation in any investigational drug study within the past 4 weeks
* No HIV-positive patients receiving antiretroviral therapy
* No concurrent CYP3A4/5 inducers or inhibitors

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib in Combination With Radiotherapy: Erlotinib (150 mg) administered orally once daily starting day 1 and continued with radiotherapy (RT) and through day 365 (one year therapy duration). RT will be administered day 1-28 (Mon-Fri) in dose of 1.8 Gy per fraction.
Period: Overall Study
Arm/Group | Erlotinib in Combination With Radiotherapy
Started | 22
Completed | 3
Not Completed | 19
Not completed — Disease progression | 6
Not completed — Adverse Event | 4
Not completed — Patient refused | 2
Not completed — Other | 1
Not completed — Death | 1
Not completed — Not treated (became ineligible) | 4
Not completed — Not treated (changed mind) | 1

BASELINE CHARACTERISTICS:
Population: All Treated Patients
Arm/Group | Erlotinib in Combination With Radiotherapy
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.94 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib in Combination With Radiotherapy
Number analyzed (Participants) | 17
months | 7.3 [3.8 to 22.3]

2. Secondary Outcome: Complete Response
Description: Response assessment by CT scans and upper endoscopy performed between 4-8 weeks after completion of radiation.
  Complete Response (CR) is defined as absence of viable tumor in endoscopic evaluation post chemoradiation, with four-quadrant biopsies taken at 1 cm intervals throughout length of original tumor.
Time Frame: 4-8 weeks after completion of radiation.
Population: Patients Treated with Study Therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib in Combination With Radiotherapy
Number analyzed (Participants) | 17
percentage of participants | 11.76 [1.46 to 36.44]

3. Secondary Outcome: Progresssion-Free Survival
Description: Progression is defined as at least a 20% increase in the sum of long distance of target lesions taking as reference the smallest sum long distance recorded since the treatment started or the appearance of one or more new lesions, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Every 3 months, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib in Combination With Radiotherapy
Number analyzed (Participants) | 17
months | 4.5 [2.4 to 7.3]

4. Secondary Outcome: Effect of Study Therapy on Overall Quality of Life as Assessed by FACT-E Scale
Description: Functional Assessment of Cancer Therapy-Esophagus (FACT-E) is a health-related quality of life instrument validated in esophageal cancer patients. All of the scales and single-item measures range in score from 0 to 4. The ranges of average quality of life scores was from 0 to 4 and was adjusted as lower scores indicate better outcomes
Time Frame: Baseline and Week 3
Population: Patients Treated with Study Therapy and with FACT-E scores available
Measure: Median (Full Range); unit: FACT-E Score
Groups:
- Erlotinib in Combination With Radiotherapy at Baseline; Erlotinib in Combination With Radiotherapy at Week 3: Erlotinib (150 mg) administered orally once daily starting day 1 and continued with radiotherapy (RT) and through day 365 (one year therapy duration). RT will be administered day 1-28 (Mon-Fri) in dose of 1.8 Gy per fraction.
Arm/Group | Erlotinib in Combination With Radiotherapy at Baseline | Erlotinib in Combination With Radiotherapy at Week 3
Number analyzed (Participants) | 17 | 14
FACT-E Score | 1.05 [.16 to 2.61] | 1.36 [.51 to 2.26]
Statistical Analysis 1: Comparison: Erlotinib in Combination With Radiotherapy at Baseline; Test type: Superiority or Other; p = 0.011, Wilcoxon signed rank test

5. Secondary Outcome: Correlation of Smoking Status With Overall Survival
Time Frame: 5 years
Population: Patients Treated with Study Therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Current Smokers | Former Smokers | Never Smokers
Number analyzed (Participants) | 3 | 12 | 2
months | 2.4 [2.4 to 7.3] | 7.2 [3.8 to 42] | 16.6 [10.9 to 22.3]
Statistical Analysis 1: Comparison: Current Smokers vs Former Smokers vs Never Smokers; Test type: Superiority or Other; p = 0.115, Log Rank

6. Secondary Outcome: Response by Epidermal Growth Factor Receptor (EGFR) Expression
Time Frame: Radiologic evaluation every 3 months, up to 5 years
Measure: Number; unit: participants
Groups:
- EGFR<=120 μg/ml: Cut at median of 120 EGFR<=120 μg/ml
- EGFR>120 μg/ml: Cut at median of 120 EGFR>120 μg/ml
Arm/Group | EGFR<=120 μg/ml | EGFR>120 μg/ml
Number analyzed (Participants) | 8 | 8
participants
  Non-responder | 6 | 5
  Responder | 2 | 3
Statistical Analysis 1: Comparison: EGFR<=120 μg/ml vs EGFR>120 μg/ml; Test type: Superiority or Other; p = 1.000, Fisher Exact

7. Secondary Outcome: Response by Phosphor Epidermal Growth Factor Receptor (pEGFR) Expression
Time Frame: Radiologic evaluation every 3 months, up to 5 years
Measure: Number; unit: participants
Groups:
- pEGFR<=20 μg/ml: Cut at median of 20 pEGFR<=20 μg/ml
- pEGFR>20 μg/ml: Cut at median of 20 pEGFR>20 μg/ml
Arm/Group | pEGFR<=20 μg/ml | pEGFR>20 μg/ml
Number analyzed (Participants) | 8 | 8
participants
  Non-responder | 5 | 6
  Responder | 3 | 2
Statistical Analysis 1: Comparison: pEGFR<=20 μg/ml vs pEGFR>20 μg/ml; Test type: Superiority or Other; p = 1.000, Fisher Exact

8. Secondary Outcome: Response by EGFR Mutation Status
Time Frame: Radiologic evaluation every 3 months, up to 5 years
Measure: Number; unit: participants
Groups:
- No EGFR Mutation; EGFR Mutation: Assessed by fluorescent in situ hybridization (FISH)
Arm/Group | No EGFR Mutation | EGFR Mutation
Number analyzed (Participants) | 12 | 4
participants
  Nonresponder | 9 | 2
  Responder | 3 | 2
Statistical Analysis 1: Comparison: No EGFR Mutation vs EGFR Mutation; Test type: Superiority or Other; p = 0.5467, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Erlotinib in Combination With Radiotherapy
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib in Combination With Radiotherapy (N=17)
Cardiac failure congestive - Grade 5 (Cardiac disorders) | 1 (1)
Myocardial infarction - Grade 4 (Cardiac disorders) | 1 (1)
Diarrhoea - Grade 3 (Gastrointestinal disorders) | 3 (5)
Ileus - Grade 3 (Gastrointestinal disorders) | 2 (2)
Oesophageal stenosis - Grade 2 (Gastrointestinal disorders) | 1 (1)
Death - Grade 5 (General disorders) | 2 (2)
Fatigue - Grade 3 (General disorders) | 1 (1)
Non-cardiac chest pain - Grade 3 (General disorders) | 1 (1)
Pneumonia - Grade 3 (Infections and infestations) | 1 (1)
Haemoglobin - Grade 2 (Investigations) | 1 (1)
Dehydration - Grade 3 (Metabolism and nutrition disorders) | 3 (4)
Hyperglycaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorder - Grade 4 (Nervous system disorders) | 1 (1)
Dyspnoea - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib in Combination With Radiotherapy (N=17)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 1 (2)
Anaemia - Grade 2 (Blood and lymphatic system disorders) | 2 (2)
Leukopenia - Grade 1 (Blood and lymphatic system disorders) | 3 (4)
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia - Grade 1 (Blood and lymphatic system disorders) | 7 (10)
Lymphopenia - Grade 2 (Blood and lymphatic system disorders) | 11 (17)
Lymphopenia - Grade 3 (Blood and lymphatic system disorders) | 8 (10)
Lymphopenia - Grade 4 (Blood and lymphatic system disorders) | 2 (2)
Neutropenia - Grade 1 (Blood and lymphatic system disorders) | 1 (2)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Acute myocardial infarction - Grade 4 (Cardiac disorders) | 1 (1)
Angina pectoris - Grade 1 (Cardiac disorders) | 1 (1)
Angina pectoris - Grade 2 (Cardiac disorders) | 1 (2)
Ventricular arrhythmia - Grade 4 (Cardiac disorders) | 1 (1)
Vision blurred - Grade 3 (Eye disorders) | 1 (1)
Abdominal distension - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 3 (3)
Chapped lips - Grade 1 (Gastrointestinal disorders) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 2 (2)
Constipation - Grade 2 (Gastrointestinal disorders) | 1 (2)
Diarrhoea - Grade 1 (Gastrointestinal disorders) | 8 (16)
Diarrhoea - Grade 2 (Gastrointestinal disorders) | 3 (3)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Dyspepsia - Grade 2 (Gastrointestinal disorders) | 1 (1)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 2 (2)
Dysphagia - Grade 2 (Gastrointestinal disorders) | 5 (5)
Dysphagia - Grade 3 (Gastrointestinal disorders) | 2 (2)
Eructation - Grade 1 (Gastrointestinal disorders) | 1 (1)
Flatulence - Grade 1 (Gastrointestinal disorders) | 1 (1)
Gastritis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease - Grade 1 (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying - Grade 2 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 6 (10)
Nausea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 3 (Gastrointestinal disorders) | 1 (1)
Odynophagia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Odynophagia - Grade 2 (Gastrointestinal disorders) | 1 (1)
Oesophageal obstruction - Grade 3 (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis - Grade 2 (Gastrointestinal disorders) | 2 (2)
Oesophageal stenosis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Oesophagitis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Oesophagitis - Grade 2 (Gastrointestinal disorders) | 2 (2)
Reflux oesophagitis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis - Grade 2 (Gastrointestinal disorders) | 2 (2)
Retching - Grade 1 (Gastrointestinal disorders) | 1 (1)
Stomatitis - Grade 1 (Gastrointestinal disorders) | 2 (2)
Stomatitis - Grade 2 (Gastrointestinal disorders) | 2 (2)
Vomiting - Grade 1 (Gastrointestinal disorders) | 4 (8)
Vomiting - Grade 2 (Gastrointestinal disorders) | 3 (3)
Chills - Grade 1 (General disorders) | 1 (1)
Early satiety - Grade 2 (General disorders) | 1 (1)
Fatigue - Grade 1 (General disorders) | 11 (14)
Fatigue - Grade 2 (General disorders) | 12 (12)
Fatigue - Grade 3 (General disorders) | 1 (1)
Mucosal inflammation - Grade 1 (General disorders) | 4 (6)
Oedema - Grade 1 (General disorders) | 1 (1)
Oedema peripheral - Grade 1 (General disorders) | 3 (3)
Oedema peripheral - Grade 2 (General disorders) | 1 (1)
Pain - Grade 2 (General disorders) | 3 (3)
Hyperbilirubinaemia - Grade 1 (Hepatobiliary disorders) | 2 (4)
Hyperbilirubinaemia - Grade 2 (Hepatobiliary disorders) | 1 (1)
Fungal skin infection - Grade 1 (Infections and infestations) | 1 (1)
Fungal skin infection - Grade 2 (Infections and infestations) | 1 (2)
Infection - Grade 2 (Infections and infestations) | 1 (2)
Urinary tract infection - Grade 2 (Infections and infestations) | 2 (2)
Contusion - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Procedural site reaction - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased - Grade 1 (Investigations) | 3 (3)
Aspartate aminotransferase - Grade 1 (Investigations) | 2 (2)
Aspartate aminotransferase increased - Grade 1 (Investigations) | 5 (7)
Aspartate aminotransferase increased - Grade 2 (Investigations) | 1 (1)
Blood alkaline phosphatase - Grade 1 (Investigations) | 2 (3)
Blood alkaline phosphatase - Grade 2 (Investigations) | 1 (1)
Blood alkaline phosphatase increased - Grade 1 (Investigations) | 1 (1)
Blood bilirubin - Grade 1 (Investigations) | 2 (2)
Blood bilirubin - Grade 2 (Investigations) | 2 (2)
Blood bilirubin increased - Grade 1 (Investigations) | 1 (1)
Blood bilirubin increased - Grade 2 (Investigations) | 1 (2)
Blood calcium decreased - Grade 1 (Investigations) | 1 (1)
Blood creatine - Grade 2 (Investigations) | 1 (1)
Blood creatine increased - Grade 1 (Investigations) | 1 (1)
Blood creatinine - Grade 1 (Investigations) | 3 (3)
Blood creatinine - Grade 2 (Investigations) | 1 (5)
Haemoglobin - Grade 1 (Investigations) | 6 (7)
International normalised ratio increased - Grade 1 (Investigations) | 1 (1)
International normalised ratio increased - Grade 2 (Investigations) | 1 (1)
International normalised ratio increased - Grade 3 (Investigations) | 1 (2)
Platelet count decreased - Grade 1 (Investigations) | 4 (6)
Troponin I increased - Grade 4 (Investigations) | 1 (1)
Weight decreased - Grade 1 (Investigations) | 10 (11)
Weight decreased - Grade 2 (Investigations) | 5 (5)
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 4 (6)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 5 (6)
Anorexia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Dehydration - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Dehydration - Grade 2 (Metabolism and nutrition disorders) | 5 (6)
Gout - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia - Grade 1 (Metabolism and nutrition disorders) | 4 (7)
Hyperglycaemia - Grade 2 (Metabolism and nutrition disorders) | 4 (5)
Hyperkalaemia - Grade 1 (Metabolism and nutrition disorders) | 3 (4)
Hypernatraemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 4 (6)
Hypocalcaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (4)
Hypocalcaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia - Grade 1 (Metabolism and nutrition disorders) | 6 (8)
Hyponatraemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Arthralgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3)
Buttock pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Gouty arthritis - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness - Grade 1 (Nervous system disorders) | 1 (3)
Dizziness - Grade 2 (Nervous system disorders) | 1 (1)
Dysgeusia - Grade 1 (Nervous system disorders) | 4 (5)
Headache - Grade 1 (Nervous system disorders) | 1 (1)
Syncope - Grade 3 (Nervous system disorders) | 2 (2)
Tremor - Grade 1 (Nervous system disorders) | 1 (1)
Depression - Grade 1 (Psychiatric disorders) | 1 (1)
Depression - Grade 2 (Psychiatric disorders) | 2 (2)
Insomnia - Grade 1 (Psychiatric disorders) | 1 (1)
Insomnia - Grade 2 (Psychiatric disorders) | 2 (2)
Pollakiuria - Grade 2 (Renal and urinary disorders) | 1 (1)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dysphonia - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
Drug eruption - Grade 2 (Skin and subcutaneous tissue disorders) | 3 (4)
Hyperhidrosis - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (4)
Palmar-plantar erythrodysaesthesia syndrome - Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 6 (14)
Rash - Grade 2 (Skin and subcutaneous tissue disorders) | 7 (8)
Rash pruritic - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis - Grade 3 (Vascular disorders) | 1 (1)
Hypotension - Grade 2 (Vascular disorders) | 1 (1)
Hypotension - Grade 4 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 1 (Vascular disorders) | 1 (2)
Orthostatic hypotension - Grade 2 (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes